CLINICAL TRIAL: NCT03717272
Title: A Phase 2, Single Center, Double-Blind, Placebo-Controlled, Randomized, Dose-Ranging Cross Over Study to Evaluate the Effects of Multiple Oral Doses of AEF0117 on the Subjective Effects of Cannabis and Cannabis Self-Administration in Subjects With CUD
Brief Title: Effect of AEF0117 on Subjective Effects of Cannabis in CUD Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other); New York State Psychiatric Institute (Other); ClinStar, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AEF0117-201; 5R01DA038875-02 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2018-10-24 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Marijuana Abuse
Keywords: AEF0117; Cannabis-related Use Disorder; Cannabis subjective effects; Cannabis self-administration; cannabis-induced analgesia; cannabis-related cognitive disorder
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AEF0117 (Experimental): AEF0117 capsules ; dose range 0.02 to 1.2mg by mouth, once a day for 5 consecutive days.
  Interventions: Drug: AEF0117; Drug: Placebo oral capsule
- Placebo oral capsule (Placebo Comparator): corn oil capsules once a day for 5 consecutive days.
  Interventions: Drug: AEF0117; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: AEF0117 — AEF0117 capsules
Drug: Placebo oral capsule — Corn oil capsule manufactured to mimic AEF0117 capsule

SUMMARY:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. Approximately 9 % of those who use cannabis will become addicted. The number goes up to about 1 in 6 among those who start using cannabis as teenagers and to 25 to 50 % among those who smoke cannabis daily. The consequences of cannabis abuse in the most prone population (14-25 years of age) are extremely serious, and may include addiction, altered brain development, poorer educational outcomes, cognitive impairment, lower income, greater welfare dependence, unemployment and lower relationship and life satisfaction. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET (Administration, Distribution, Metabolism, Elimination and Toxicology) in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders. The purpose of this research is to study how AEF0117 influences the subjective effects of cannabis in subjects with CUD. AEF0117 acts in the same parts of the brain as THC (tetrahydrocannabinol), the active ingredient of marijuana, and may temporarily alter some of cannabis's effects.

This will be a single center study in healthy male and non-pregnant female, non-treatment seeking, cannabis smoking subjects with cannabis use disorder (CUD). The study design will be a randomized, double-blind, placebo-controlled, cross-over design, multiple dose escalation study with AEF0117. This study is designed to test the effects of two to four doses of AEF0117 compared to placebo on primarily peak subjective effects of cannabis as primary objectives. The secondary objectives are to test the effects of AEF0117 compared to placebo on cannabis self-administration, on cannabis-induced analgesia and on cognitive performance in cannabis smoking subjects. The study hypothesis is that AEF0117 will decrease ratings of cannabis' positive subject effects (e.g., 'good drug effect', high) and decrease cannabis self-administration compared to placebo and also decrease the other unconditioned effects of cannabis studied here. Each subject will have a screening visit, then be included for two 6-day inpatient periods separated by a minimum 14-day outpatient washout. Subjects will be advised that they will receive both active and placebo study medication but will remain blinded to whether they will receive AEF0117 or placebo on Period A and Period B. Each period is composed of 5 consecutive days of treatment (active or placebo), one administration per day. Research staff that interacts with study subjects will also remain blinded to whether subjects are receiving AEF0117 or placebo. The study duration for the first 3 doses of AEF0117 is estimated to be approximately up to 10 months from the start of subject recruitment to the last subject last visit.

DETAILED DESCRIPTION:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. Approximately 9 % of those who use cannabis will become addicted. The number goes up to about 1 in 6 among those who start using cannabis as teenagers and to 25 to 50 % among those who smoke cannabis daily. The consequences of cannabis abuse in the most prone population (14-25 years of age) are extremely serious, and may include addiction, altered brain development, poorer educational outcomes, cognitive impairment, lower income, greater welfare dependence, unemployment and lower relationship and life satisfaction. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders. The purpose of this research is to study how AEF0117 influences the subjective effects of cannabis in subjects with CUD. AEF0117 acts in the same parts of the brain as THC, the active ingredient of marijuana, and may temporarily alter some of cannabis's effects.

This will be a single center study in healthy male and non-pregnant female, non-treatment seeking, cannabis smoking subjects with cannabis use disorder (CUD). The study design will be a randomized, double-blind, placebo-controlled, cross-over design, multiple dose escalation study with AEF0117. This study is designed to test the effects of two to four doses of AEF0117 compared to placebo on primarily peak subjective effects of cannabis as primary objectives. The secondary objectives are to test the effects of AEF0117 compared to placebo on cannabis self-administration, on cannabis-induced analgesia and on cognitive performance in cannabis smoking subjects. The study hypothesis is that AEF0117 will decrease ratings of cannabis' positive subject effects (e.g., 'good drug effect', high) and decrease cannabis self-administration compared to placebo and also decrease the other unconditioned effects of cannabis studied here. It is hypothesized that AEF0117 will antagonize cannabis effects on the basis of data: (a) in mice showing that AEF0117 antagonized all unconditioned effects of THC tested; (b) in rats showing that AEF0117 decreased THC- induced dopamine release, and (c) in nonhuman primates showing that AEF0117 antagonized THC self-administration and THC-induced reinstatement of THC seeking. The study is also designed to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of escalating multiple oral doses of AEF0117 in adult male and non-pregnant female, nontreatment seeking, cannabis smoking subjects with cannabis use disorder (CUD). In this study, subjects will be closely monitored through adverse event monitoring and vital signs measurements. This study will be conducted in adherence to the study protocol, Good Clinical Practices (GCP). Data from this study will be used to aid the design of future clinical studies in patients.

This protocol represents the first clinical study of AEF0117 in subjects with cannabis use disorder and the third clinical study of AEF0117 in humans, therefore, the risks and benefits in this patient population are not well known. The study hypothesis is that AEF0117 will not precipitate withdrawal in cannabis abusers at any of the doses tested because (a): its signaling-specific effects only partially modify the activity of the CB1 (cannabinoid receptor type 1) receptor, and (b) AEF0117 did not precipitate withdrawal in THC-dependent mice at doses 30 times higher than the ED50 (median effective dose ) antagonizing most of the behavioral effects of THC.

This will be a single-center study conducted in the USA. Approximately 48 cannabis-smoking subjects with cannabis use disorder will be randomized into the study for the first 3 doses of AEF0117. 16 additional cannabis-smoking subjects with CUD could be randomized into the study for completion of Cohort 4. The study duration for the first 3 doses of AEF0117 is estimated to be up to 10 months from the start of subject recruitment to the last subject last visit. Each subject will have a screening visit, then be included for two 6-day inpatient periods separated by a minimum 14-day outpatient washout period. Subjects will provide signed informed consent upon enrollment into the study. Subjects will be advised that they will receive both active and placebo study medication but will remain blinded to whether they will receive AEF0117 or placebo in Period A and Period B. Each period is composed of 5 consecutive days of treatment (active or placebo), one administration per day. Research staff who interact with study subjects will also remain blinded as to whether subjects are receiving AEF0117 or placebo.

At least two multiple oral doses of AEF0117 will be tested in order to establish a dose response of AEF0117 effects. The anticipated target dose is 0.2mg (referred to as 1x dose). The starting dose will be 0.06 mg corresponding to the 0.3x dose. The anticipated doses range will range between 0.02 and 1.2 mg that are respectively the 0.1x and the 6x dose levels. The 30x dose level has been evaluated in phase 1 studies in healthy volunteers with demonstration of good safety and tolerability even at this supratherapeutic dose level. At the end of each cohort, available efficacy, safety and tolerability data will be reviewed for all subjects as a function of active (AEF0117) versus placebo medication by a data monitoring consortium consisting of the principal investigator, the sponsor and external representatives of a Data Safety Monitoring Board (DSMB). The above representatives will receive an unblinded interim report on these data (Safety and Efficacy Interim Report) and they will only be unblinded to data from the finalized cohort. The doses administered in cohort 2 and cohort 3 will be decided according to the decision process summarized below:

First cohort dose: 0.06mg (0.3x dose) Second Cohort dose will be either: a. 0.2mg (1x dose) if the 0.06 mg dose induces a decrease < 70% in cannabis subjective effects; or b. 0.02 mg (0.1x dose) if the 0.06 mg dose induces a reduction >70% in cannabis subjective effects.

Third cohort dose if second cohort dose = 0. 2 mg then the dose will be either: a. 0.6mg (3x dose) if 0.2 and 0.06 mg doses do not induce a significant reduction in cannabis subjective effects; or b. 0.6 mg if the reduction in cannabis subjective effects at 0.2mg is > to the one at 0.06 mg; or c. 0.02 mg if the reduction induced by 0.06mg is ≤ a significant reduction induced by 0.2 mg. Third cohort dose if second cohort dose = 0.02 mg: then the dose will be 0.2 mg (1x dose) if the reduction induced by 0.02mg is ≤ the reduction induced by 0.06 mg.

Fourth cohort dose if third cohort dose = 0. 6 mg then the dose will be: a. 1.2mg (6x dose) if 0.06, 0.2 and 0.6 do not induce a significant reduction in cannabis subjective effects; or b. 1.2 mg if the reduction in cannabis subjective effects at 0.6mg is > to the one at 0.2 mg.

The planned dose escalation schema may be amended based on the ongoing safety and efficacy data.

Each dose will be tested in an independent cohort of subjects (estimated inclusion of up to n=16 per dose). Subjects will be recruited in group of 4 subjects until n=12 have completed each dose cohort to ensure that there is sufficient statistical power to analyze the efficacy of AEF0117 in attenuating cannabis subjective effects (e.g., good drug effect, high).

For both periods of treatment (A and B), eligible subjects will be admitted to the research center by approximately 1200 h in the afternoon prior to Day 1 and will remain confined at the research facility until the morning of Day 6. Subjects randomized to Group 1 will receive AEF0117 in Period A and placebo in Period B. Subjects randomized to Group 2 will receive placebo in Period A and AEF0117 in Period B. According to the pharmacokinetic properties of AEF0117 extrapolated from the pharmacokinetic results of the previous phase I studies (AEF0117 101 and AEF0117-102), a minimum of 14 days of washout will be scheduled between Period A and Period B.

Subjects will be awakened at approximately 0800 h on study days, will receive food boxes, will have vital sign measurements (sitting blood pressure, pulse rate, weight) and will complete a subjective-effects and a sleep questionnaire. Study medication containing either AEF0117 or placebo will be administered at approximately 0900 h on Days 1-5 of both period A and period B.

Plasma samples for PK and PD (except cortisol, estradiol and progesterone) analysis will be obtained at predose, 3 h, 9.5 h and 24 h after the first administration and at Day 6 (24 h after the last administration on Day 5) of each period. Cortisol, estradiol and progesterone analysis will be obtained at predose on Day1 and on Day6 (at 24h after the last administration on Day5) of both periods.

On each Study Day, at approximately 1230 h, subjects will receive an experimenter-administered 'sample' of 6 puffs of cannabis (1 5-second puff/minute). Then at 1250 h, 1310 h, 1330 h, 1400 h and 1415 h, subjects will complete a subjective-effects questionnaire and a cannabis rating form. At 1330 h, subjects will also complete a cognitive task battery.

On day 1, at 1430 h, subjects will receive a baseline evaluation of their pain threshold and tolerance using the CPT (cold pressor test). They will then receive at 1445 h another experimenter-administered sample of cannabis. The CPT will be repeated at 30, 60, 90, 120 and 180 min after cannabis administration.

Beginning at 1415 h on Study Days 2 through 5, subjects will be given the option to self-administer individual puffs of cannabis (up to 6 puffs/time point) every 2.0 hour until 2030 h (maximum = 24 puffs). Subjects will have to purchase the cannabis puffs using their study stipends ($2/puff).

Cannabis self-administration and food intake will be recorded and mood, sleep, cognitive and cardiovascular effects will be measured repeatedly throughout each study day Safety monitoring (vital sign measurement and adverse event monitoring) will be performed throughout the study. Subjects will have a safety evaluation on Days 6 of each Period.

Specific instruments for evaluating cannabis effects will include:

* Visual Analogue Scales (VAS) - 44-item VAS instrument which assesses mood, positive subject effects, physical symptoms, medication effects, drug craving and subjective ratings of sleep. Based on a cluster analysis, arithmetic means of individual item scores reduces the 44-items VAS into six subscales including: 'good drug effect', 'irritable', 'anxious', 'bad effect', 'tired' and 'social'. As primary endpoint, the evaluation of AEF0117 effects on peak changes in the subjective effects of cannabis (e.g. good drug effect, high) will be assessed using the "Good Drug Effect" subscale.
* Cannabis Rating Form - 5 item VAS scale which evaluates the cannabis effects that they just smoked.
* Cognitive Performance Battery -A series of 4 tasks measuring attention (Sustained Attention to Response Task), processing speed (Digit Symbol Substitution Task), recognition memory (Behavioral Pattern Separation Task) and Reaction Time/Response Inhibition (Color Stroop).
* Objective Sleep Measures - subjects will wear an Actiwatch® Activity Monitoring System that records objective sleep outcomes (e.g., sleep latency, sleep efficiency).
* Sleep questionnaire - 7-item VAS instrument that assesses the quality of sleep and how many hours slept the previous night and wakefulness in the morning on Study Days 1-6.
* Cardiovascular effects - sitting heart rate and blood pressure are measured at 0830 h (baseline i.e., predose) and at 1200 h (3 hours post medication administration). A blood pressure cuff will be placed on the non-dominant arm with connections to a Sentry II automated vital signs monitor.
* Food intake - a wide range of food items will be available ad libitum to subjects throughout each study day. Restrictions on foods include grapefruits, Seville oranges, tangelos, grapefruit, orange and apple juices. Daily caloric intake will be calculated (subject's daily recording of time and quantity of food consumed will be verified by an examination of food trash).

Adverse events will be monitored by research staff and medical observations and spontaneous reporting throughout the study. The grading system of adverse events used in this study will be the grading system proposed by Sibille M., et. al. Specifications on the grading system for clinical observations and ECG parameters will be based on the publication by Sibille M, Patat A, et al. Vital signs and laboratory parameters will be based on the FDA vaccine guidance (The Biologics Blood Vaccines Guidance Compliance, FDA). The planned dosing escalation schedule can be modified during the course of the study based on the efficacy and safety data. At the end of each cohort, efficacy and safety data of each cohort from Day 1 through to the morning of Day 6 of each Period will be evaluated in all subjects in this cohort as a function of active (AEF0117) versus placebo medication by a data monitoring consortium consisting of the principal investigator, the sponsor and external representatives of a Data Safety Monitoring Board (DSMB). The above representatives will receive an unblinded interim report on these data and they will only be unblinded to data from the finalized cohort. Interim reports prepared for the evaluation of the dose escalation will be made and the decision to progress to the next dose or to modify the subsequent dose will be jointly made by the principal investigator, the sponsor and the external representatives of the DSMB according to a predefined charter. The planned dose escalation may be modified to include the repetition of a dose, to escalate to an intermediate dose level (i.e., to a higher or lower increment of dose).

However, dose escalation and dose administration within the same cohort should discontinue if at least one of the drug related stopping criteria described below is observed within the same cohort.

* Criterion 1: Occurrence of any serious (grade 4) adverse event (SAE).
* Criterion 2: Occurrence of any severe (grade 3) adverse events (AE) in 2 or more subjects treated with AEF0117 at any given dose (evaluated after un-blinding during the study).

In the event criterion 1 or 2 is reached, the dose escalation will be discontinued, unless the AE is determined by the Investigator, the Sponsor and the external representatives of the DSMB to be clearly unrelated to the administration of the study medication and has a clear alternative explanation.

* Criterion 3: Moderate (grade 2) adverse events (AE's) is at least a safety alert leading to cautious and closer assessment of safety in other subjects. An upgrading applies if rapid worsening, concomitant laboratory findings, clinical symptoms and signs occur.
* Criterion 4: Changes in clinical signs grade 2 of the same character (similar abnormality) in 3 or more subjects.
* Criterion 5: Changes in vital signs grade 2 of the same character (similar abnormality) in 3 or more subjects.

In the event criteria 3, 4 and 5 are reached, the dose escalation scheme may be modified by repeating the dose, by lowering the dose or decreasing the increment of dose escalation and continue the study with a new cohort of subjects.

Although these are the minimum criteria, dose escalation may be suspended on the basis of other safety information considered to pose a risk to the subjects and agreed to between the sponsor and the investigator. The number of subjects evaluated for pharmacodynamic endpoints and safety assessments for dose escalation determination (i.e., 12-16 subjects at each dose level) is empirically based and not based on a formal sample size determination.

A sample size of 12 completers will provide at least 90% statistical power to detect changes in subjective effects as a function of medication. Based on treatment effects and variability observed in an earlier study and the hypothesis that AEF0117 will decrease ratings of cannabis' positive subjective effects (e.g., 'good drug effect'; high), a sample size of 12 would have a 90% power for detecting a mean difference of 36 mm on a 100 mm VAS scale in a cross-over design at p = 0.05 (two-tailed).

Mood, physical symptoms, food intake, sleep, cognitive task performance, and cardiovascular effects will be analyzed using repeated measures analysis of variance (ANOVA) models. A cluster analysis of peak subjective-effects ratings to reduce the overall number of comparisons will be employed. Tests of differences will be based on F statistics with degrees of freedom corrected, depending on the observed within-subject correlation of the measures, using the method of Huynh and Feldt. Planned contrasts will be single degree of freedom comparisons using the appropriate interaction error term. Results will be considered statistically significant at p < 0.05, using 2-tailed tests.

Repeated-measures analysis of variance will be used to assess cannabis's peak analgesic effects as a function of medication condition (active or placebo AEF0117). Dependent variables will include pain sensitivity and tolerance and subjective pain effects as assessed by the pain intensity and bothersomeness scales. For each medication condition, pain sensitivity and tolerance will be calculated for each participant as the percent of the baseline pre-dosing CPT response. Results will be considered statistically significant when p-values are equal to or less than 0.05 using Huynh-Feldt corrections.

Plasma pregnenolone, DHEA (dehydroepiandrosterone ), testosterone, allopregnanolone, endocannabinoids (AEA and 2AG), concentrations will be summarized for AEF0117 and placebo using descriptive statistics. Serum cortisol, estradiol and progesterone concentrations will be summarized for AEF0117 and placebo using descriptive statistics. Pharmacokinetic Analyses:

Plasma AEF0117, THC and the metabolites 11-OH-THC (11-hydroxy-THC) and 11-COOH-THC (11-carboxy-THC) concentrations will be summarized descriptively by dose and displayed graphically.

Safety evaluations (adverse events monitoring, vital signs measurements and appearance of signs of cannabis withdrawal) will be summarized for AEF0117 and placebo by dose level and pooled doses using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male, at least 21 years old and no more than 60 years old, inclusively. As the effect of the study drug on sperm is still unknown, male subjects will be instructed to refrain from donating sperm or planning a pregnancy during the study and for 90 days after study completion. They will be instructed to tell the study doctor if their partner becomes pregnant during the study or during 90 days after study completion. Male subjects will have to use double-barrier contraceptive methods: male condoms and spermicide.
* Be a healthy, non-pregnant female, at least 21 years old and no more than 60 years old, inclusively, and meet one of the following criteria with regard to child-bearing status:

  1. Be a woman of non-child-bearing potential, defined as surgically sterile (e.g., hysterectomy, tubal ligation) or post-menopausal [amenorrhea >1 year and FSH (follicle stimulating hormone) > 30 microU/ml] with a negative pregnancy test; OR
  2. Be a woman of child-bearing potential and practicing a highly effective method of contraception (i.e., >99% effective when used consistently and correctly, or, in other words, <1% failure rate per year) including the following methods: Intrauterine Copper Contraceptive (as for example, Paragard T 380A), sexual abstinence, or vasectomized male partner with a negative pregnancy test.
* Have a body mass index (BMI) within the range of >18.5 and <32 kg/m2 unless approved by the sponsor and investigator.
* Be a current cannabis smoker of ≥ 1 grams of cannabis per day, at least 6 days per week.
* Meet the diagnostic criteria for Cannabis Use Disorder (CUD) based on DSM-5 criteria
* Have no significant diseases in their medical history or clinically significant findings on physical examination or clinical laboratory evaluations.
* Be informed of the nature of the study and provide signed informed consent.
* Be legally competent and able to communicate effectively with study personnel.

Exclusion Criteria:

* Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems.
* The presence of clinically significant laboratory values. Subjects with AST (aspartate aminotransferase), ALT (alanine transaminase) or GGT (gamma-glutamyltransferase) values >2x the upper limit of normal, alkaline phosphatase, bilirubin, BUN (blood urea nitrogen), creatinine >15% above the upper limit of normal, or hemoglobin or hematocrit level >15% below the lower limit of normal may only be enrolled upon joint agreement of the sponsor and investigator.
* Have abnormal baseline values for the steroid hormones: cortisol, testosterone, estradiol and progesterone in accordance to their reproductive status (for example but not limited to surgical or post-menopausal).
* A history of alcoholism or drug addiction other than cannabis use disorder within the past 2 years, or positive results from a urine screen for substances of abuse other than THC.
* A history of smoking greater than 20 cigarettes per day on average, in the month prior to Screening, or having an inability to abstain from smoking (or use of any nicotine-containing substance) for at least 8 hours.
* A history of major Axis I psychopathology, e.g., mood disorder with functional impairment, schizophrenia).
* Inadequate venous access.
* A known history of Hepatitis B or C or HIV infection.
* Ingestion of an investigational drug or product, or participation in a drug study within a period of 30 days prior to screening (for investigational drugs with an elimination half-life greater than 10 days, this will be extended to 60 days).
* Use of any prescription or over-the-counter (OTC) drug therapy, including herbal, homeopathic, vitamins, minerals and nutritional supplements, unapproved by the sponsor, within 2 weeks prior to receiving the study medication (for drugs with an elimination half-life greater than 10 days, this will be extended to 60 days). The use of any food supplement or body cream containing pregnenolone or any other steroid including phytosteroids.
* Use of a drug therapy known to induce or inhibit hepatic drug metabolism within 30 days prior to screening or during the study.
* Unable to follow the restrictions outlined in the protocol.
* Previous participation in a cohort for any dose level of AEF0117.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Subjective Effects of Cannabis | On Days 1, 2, 3, 4 and 5 of each Period: Mean VAS will be assessed predose and postdose
  Mean Visual Analog Scale (VAS) rating assessing positive subjective drug effect, (Good Drug Effect). This scale uses a 0-100mm rating, where higher numbers indicate a better drug effect.

SECONDARY OUTCOMES:
Changes in cannabis self-administration | On Days 2, 3, 4 and 5 of each Period: at 5.5 hours, 7.5 hours , 9.5 hours and 11.5 hours post dose
  Number of purchased puffs of cannabis cigarette per day (possibility of 0-24 puffs per day). Higher numbers indicate more cannabis self-administration.
Percent Change in Subjective Ratings of Cannabis. | On Days 1, 2, 3, 4 and 5 of each Period: CRF will be completed at 3.84 hours, 4.17 hours , 4.5 hours, 5.0 hours and 5.25 hours postdose
  Five-item Cannabis Rating Form Visual Analog Scale (CRF-VAS) where subjects report, on a 0-100mm scale, ratings of 'cannabis strength', 'liking', 'desire to take again', 'good cannabis effect', and 'bad cannabis effect'. Higher reported ratings indicate more agreement with each term.
Changes in pain threshold and pain tolerance | Baseline at 1430 hours; experimenter-administered cannabis at 1445 hours; CPT at 1515 hours, 1545 hours, 1615 hours, 1645 hours and 1745 hours
  Changes in pain response (threshold and tolerance) as a function of cannabis and medication condition will be assessed using the Cold pressor test. Pain threshold is determined by latency (in seconds) to first self-report of subjective feelings of pain while the hand is immersed in cold water (4 degrees celsius), and pain tolerance is determined by latency (in seconds) to hand withdrawal from cold water.
Cognitive Performance (Sustained Attention) | On Days 1, 2, 3, 4 and 5 of each Period, at 0.5 hours and 4.5 hours post dose
  Sustained Attention to Response Task (SART). Participants are presented with a single digit 1-9 in the middle of the screen in varying font sizes. The digit disappears after a short while and is replaced with a mask (circle with an X). Participants are asked to press the spacebar if any digit other than 3 is presented and to withhold the response if digit 3 presented. The outcome is the total number of correct suppressions. More correct suppressions indicate better cognitive performance.
Cognitive Performance (Processing speed) | On Days 1, 2, 3, 4 and 5 of each Period, at 0.5 hours and 4.5 hours post dose
  Digit Symbol Substitution Task (DSST). Participants are presented with an 18 (columns) x 16 (rows) matrix. Odd rows contain symbols, even rows contain empty answer boxes (18x8 = 144). The task is to translate the symbols into digits with the help of a provided key within a 2 min time frame. The outcome is the total number of correct responses. More correct responses indicate better cognitive performance.
Cognitive Performance (Recognition Memory) | On Days 1, 2, 3, 4 and 5 of each Period, at 0.5 hours and 4.5 hours post dose
  Behavioral Pattern Separation Task. The first part of the experiment presents 128 pictures (default) of everyday items and participants have to decide whether the item is an OUTDOOR or an INDOOR item. The second part of the experiment presents 64 of the previously seen pictures (targets), 64 of very similar items (lures), and 64 new items (foils). Participants are asked to categorize the items as old, new, or similar within 2.5s (default) The outcome is percent correct. Higher percentage correct indicates better cognitive performance.
Cognitive Performance (Reaction time) | On Days 1, 2, 3, 4 and 5 of each Period, at 0.5 hours and 4.5 hours post dose
  Color Stroop Task. Participants are given names of color words written in varying color ink, and are asked to indicate the printed color of the word (not its meaning) by pressing a key as fast as they can without making too many errors. The outcome is mean reaction time of correctly answered trials. More correctly answered trials indicates better cognitive performance.
AUC (area under curve) of AEF0117 Plasma exposure | Pharmacokinetic measures (e.g., 0, 3 hours, 9.5 hours and 24hours post first dose and 24 hours after the last dose administered on Day5
  Plasmatic exposure to AEF0117
AUC of Plasma concentrations of THC | Pharmacokinetic measures (e.g., 0, 3 hours, 9.5 hours and 24 hours post first dose and 24 hours after the last dose administered on Day5
  Plasmatic exposure to THC
AUC of Plasma concentrations of 11-OH-THC | Pharmacokinetic measures (e.g., 0, 3 hours, 9.5 hours and 24hours post first dose and 24 hours after the last dose administered on Day5
  Plasmatic exposure to 11-OH-THC
AUC of Plasma concentrations of 11-COOH-THC | Pharmacokinetic measures (e.g., 0, 3 hours, 9.5 hours and 24 hours post first dose and 24 hours after the last dose administered on Day5
  Plasmatic exposure to 11-COOH-THC
Food intake | Daily from Day 1 to Day 5 of each period
  Daily caloric intake will be calculated by recording and summing the calorie counts for all food items each participant consumes on each day. Consumption of food items will be self-reported by each participant, and verified by checking each participant's trash every day during the inpatient phase.
Sleep Quality | Each day during inpatient phase at -0.75h prior to medication dosing.
  Self-reported 7-item Visual Analog Scale (VAS) of sleep quality. Participants rate, on a 0-100mm scale, the following: 'I slept well last night', 'I woke up early this morning', 'I fell asleep easily last night', 'I feel clear-headed this morning', 'I woke up often last night', 'I am satisfied with my sleep last night', and 'I had a lot of dreams last night'. Higher ratings indicate more agreement with each statement.
Sleep Quantity | Daily from Day 1 to Day 5 of each period
  Number of hours slept as measured by an Actiwatch worn by the participant each night. Higher numbers indicate more hours slept.
Incidence of Treatment-Emergent Adverse Events [safety and tolerability] | Screening, Predose on Day 1 and on Day 6
  Collection of AE, weight, hematology, serum chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Margareth Haney, PhD, Principal Investigator — Substance Use Research Center
Locations (1):
- Substance Use Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haney M, Vallee M, Fabre S, Collins Reed S, Zanese M, Campistron G, Arout CA, Foltin RW, Cooper ZD, Kearney-Ramos T, Metna M, Justinova Z, Schindler C, Hebert-Chatelain E, Bellocchio L, Cathala A, Bari A, Serrat R, Finlay DB, Caraci F, Redon B, Martin-Garcia E, Busquets-Garcia A, Matias I, Levin FR, Felpin FX, Simon N, Cota D, Spampinato U, Maldonado R, Shaham Y, Glass M, Thomsen LL, Mengel H, Marsicano G, Monlezun S, Revest JM, Piazza PV. Signaling-specific inhibition of the CB1 receptor for cannabis use disorder: phase 1 and phase 2a randomized trials. Nat Med. 2023 Jun;29(6):1487-1499. doi: 10.1038/s41591-023-02381-w. Epub 2023 Jun 8. PMID 37291212